CLINICAL TRIAL: NCT02047916
Title: NeoAdapt 1: A Study of Circulatory Adaptation of Newborn Infants After Birth
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Dr Liam Mahoney, Clinical Research Fellow in Paediatrics, Brighton & Sussex Medical School
Other Study IDs: IRAS 145159
Record Dates: First submitted 2014-01-27; First posted 2014-01-28 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Circulatory Failure in Newborn Infants
Keywords: Neonates; Superior Vena Cava Flow; Pleth variabilty index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Neonates > 33 weeks gestation: * Neonates >33 weeks gestational age
  * Postnatal age <72 hours;
  * Parental informed consent;
  * Inpatient at the Royal Sussex County Hospital (RCSH): either receiving special care on the Trevor Mann Baby Unit (TMBU) or normal care on the postnatal ward

SUMMARY:
The current definitions of neonatal shock/circulatory failure are outdated and inaccurate. This makes the development of evidence based protocols for its treatment very difficult. Furthermore these definitions often rely on invasive methods of monitoring in patients such as an arterial line. Since the advent of functional echocardiography in neonatology there has been increased interest in non-invasive measurements of neonatal circulatory failure. However research in this field has been confined to premature infants.

The purpose of the this research is to look at non invasive methods of assessing an infants circulatory status in infants older than 33 weeks gestational age in order to fill the knowledge gap here and help in the development a new definition of neonatal circulatory failure.

DETAILED DESCRIPTION:
Research has shown that the current definitions used by doctors to assess and treat infants who have a circulatory problem are inaccurate and lead to a large differences in how doctors treat this problem in babies. Treatments for circulatory problems in babies can involve the giving of medication such as adrenaline, dobutamine or dopamine. However these drugs are not licensed for use in babies and have potentially harmful side effects.

By investigating new methods of assessing a babies circulatory status we intend to help create a new definition of circulatory failure which will in turn help doctors create further studies to identify infants with circulatory failure and find the best ways of treating this condition in babies. So far research in this area has been confined to babies born at less than 33 weeks gestation. We intend to extend the knowledge in this area to infants older that 33 weeks gestation.

This is a pilot prospective observational study in babies older that 33 weeks. Infants will been considered to be from a healthy population (i.e. receiving routine care on the postnatal care or special care on the neonatal unit). Potential participants will be approached by a member of the research team and given information about the study and informed consent will be taken.

For the first three days of their lives all included infants will have two specific measurements once a day. These are known as:-

1. Superior vena cava flow assessment- This involves measuring the blood flow through one of large veins that is connected to the babies' heart using an ultrasound machine. It is a painless procedure that is well tolerated by infants.
2. Pleth variability index- This involves placing a small probe on the baby's hand or foot that will measure their oxygen levels. This will be done at the same time as the superior vena cava flow assessment is performed. Again this is a painless procedure that is well tolerated by infants.

Prior to these measurements the infants will have there blood pressure, heart rate, oxygen saturation's and capillary refill time assessed.

This assessments will be performed in addition to the routine care they receive. Infants will therefore have these measurements performed three times for the purpose of the study. If an infant is discharged by the clinical team before the third day of life then the measurements that have been performed prior to discharge will be included in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Infant >33 weeks gestational age
* Postnatal age <72 hours;
* Parental informed consent;
* Infants receiving special care on the Trevor Mann Baby Unit or well babies on the postnatal ward

Exclusion Criteria:

* Neonates considered non-viable, with a clinical decision not to provide life support
* Infants with severe congenital hydrops fetalis needing chest or peritoneal drainage before recruitment
* Infants with congenital malformations likely to affect cardiovascular adaptation. These defects include congenital diaphragmatic hernia, gastroschisis or congenital heart defects.
* Infants in whom a surgical treatment is planned within 72 hours of birth
* Infants carrying chromosomal anomalies

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Potential candidates for enrolment will be infants admitted to the postnatal ward for routine post natal care and those admitted to the Trevor Mann Baby Unit for special care. The infants will be greater than 33 weeks´ gestation, and postnatal age below 72 hours.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Superior Vena Cava Flow (SVC) | Once a day for a maximum of three days after birth
  After consent and enrolment, Echo-D assessment for SVC flow will be performed as soon as possible after birth, preferably within 12 hours of birth. Echo D assessments will be repeated every 24 hours during the first 72 hours of postnatal life, whenever possible. We anticipate that it may only be possible to perform one set of measurements on an infant consented to the study. This is because many infants receiving postnatal or special care many infants will be discharged home before the age of 72 hours.
Pleth Variability Index (PVI) | Once a day for a maximum of three days after birth
  After consent and enrolment, PVI assessments will be performed as soon as possible after birth, preferably within 12 hours of birth. PVI assessments will be repeated every 24 hours during the first 72 hours of postnatal life, whenever possible. We anticipate that it may only be possible to perform one set of measurements on an infant consented to the study. This is because many infants receiving postnatal or special care many infants will be discharged home before the age of 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Mahoney, BMBS, MRCPCH, Principal Investigator — Brighton & Sussex Medical School/Brighton & Sussex Universitys NHS Trust
Locations (1):
- Trevor Mann Baby Unit, Brighton, Sussex, United Kingdom

REFERENCES:
- See also: This is the main clinical trial the study is associated with — http://neocirculation.eu/